CLINICAL TRIAL: NCT06841822
Title: The Impact of Ultrasound-Guided Superficial and Deep Paravertebral Nerve Blocks at the Superior Costotransverse Ligament on Hemodynamics During the Induction Phase of Thoracoscopic Lung Lobectomy: A Multicenter, Double-Blind, Randomized Controlled Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nanjing First Hospital, Nanjing Medical University (Other)
Collaborators: Geriatric Hospital of Nanjing Medical University (Other); Dushu Lake Hospital Affiliated to Soochow University (Other); Huai'an First People's Hospital (Other); Yancheng First People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: KY20240924-03-KS-01; ZKX21038 (Other: Nanjing Municipal Health Commission)
Record Dates: First submitted 2025-02-11; First posted 2025-02-24 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: Thoracic Paravertebral Block; Anesthesia Induction; Hypotension on Induction

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- SCTL superficial plane block group (S group) (Experimental): The puncture needle did not break through SCTL when the ultrasound-guided thoracic paravertebral block was performed.
  Interventions: Other: SCTL superficial plane block
- SCTL deep plane block group (T group) (Placebo Comparator): SCTL was broken by a puncture needle during the ultrasound-guided thoracic paravertebral block.
  Interventions: Other: SCTL deep plane block group

INTERVENTIONS:
Other: SCTL superficial plane block — The purpose of this study was to evaluate whether thoracic paravertebral nerve block performed on superficial SCTL (puncture needle did not break SCTL) was more beneficial to maintaining hemodynamic stability during the induction period of thoracoscopic lobectomy compared with SCTL deep plane (puncture needle break SCTL). We performed an ultrasound-guided paravertebral nerve block while keeping the puncture needle did nit to break through the SCTL. In 20 patients who required CT (3D) imaging to observe drug diffusion 30min after nerve block, cold stimulation was used 30min after the procedure to assess the degree of sensory loss, including the anterior chest wall (midclavian line), lateral chest wall (posterior axillary line), and posterior chest wall (paravertebral area).
  Arms: SCTL superficial plane block group (S group)
Other: SCTL deep plane block group — Ultrasound-guided thoracic paravertebral nerve block was routinely performed. SCTL was broken by a puncture needle during the ultrasound-guided thoracic paravertebral block. In 20 patients who required CT (3D) imaging to observe drug diffusion 30min after nerve block, cold stimulation was used 30min after the procedure to assess the degree of sensory loss, including the anterior chest wall (midclavian line), lateral chest wall (posterior axillary line), and posterior chest wall (paravertebral area).
  Arms: SCTL deep plane block group (T group)

SUMMARY:
This study aims to determine whether performing a paravertebral nerve block at the superficial surface of the superior costotransverse ligament (SCTL) (without needle penetration of the SCTL) is more effective in maintaining hemodynamic stability during the induction phase of thoracoscopic lung lobectomy compared to the deep surface of the SCTL (with needle penetration of the SCTL).

This is a multicenter, double-blind, randomized controlled trial enrolling a total of 168 participants across five hospitals. To investigate the effects of different nerve block methods on hemodynamics during induction, participants will be allocated to either the deep plane SCTL block group (T group) or the superficial plane SCTL block group (S group) using a stratified randomization scheme. The stratification accounts for a 40% proportion of hypertensive patients within each treatment group at each center.

Thirty minutes before surgery, patients will receive either an ultrasound-guided deep SCTL block (needle penetrating the SCTL) or a superficial SCTL block (needle not penetrating the SCTL) in the pre-anesthesia room. The target vertebral levels for the block are T4 and T6, and 20 mL of 0.375% ropivacaine hydrochloride solution will be injected slowly at each site. Researchers will document whether subpleural compression is observed on ultrasound imaging and monitor for complications such as hemothorax, pneumothorax, local hematoma, local anesthetic toxicity, epidural anesthesia, or total spinal anesthesia during the procedure.

Another investigator, blinded to the group allocation, will evaluate patients after the nerve block procedure, recording any occurrences of hemothorax, pneumothorax, local hematoma, local anesthetic toxicity, epidural block, or total spinal anesthesia. Cold sensitivity tests using the temperature method will be conducted at the midaxillary line within the corresponding blocked regions at 5, 10, 20, and 30 minutes post-block, and the sensory blockade level will be recorded.

Thirty minutes after the block, anesthesia induction will be performed using target-controlled infusion (TCI) of propofol and remifentanil, along with rocuronium (0.6 mg/kg). Heart rate (HR), mean arterial pressure (MAP), stroke volume (SV), cardiac index (CI), and stroke volume index (SVI) will be measured every minute from induction until 5 minutes after intubation. Hypotension is defined as a MAP decrease of 20% or an absolute MAP < 65 mmHg, while severe hypotension is defined as a MAP decrease of 30% or an absolute MAP < 55 mmHg. Hemodynamic stability will be maintained using vasoactive medications as needed.

The study will record intraoperative consumption of propofol and remifentanil, anesthesia duration, intraoperative intravenous fluid volume, urine output, blood loss, and extubation time. Postoperative assessments will include resting and movement-evoked (coughing) VAS scores at 4 and 24 hours, opioid consumption within 24 hours (oxycodone usage, first demand time, number of effective and actual demands), and additional analgesic requirements. The QOR-15 score at 24 hours and puncture-related complications within 72 hours postoperatively will be documented, along with a patient satisfaction survey at 72 hours.

For the imaging study evaluating drug diffusion following each block method using CT (3D) imaging, 40 patients will be recruited at Nanjing First Hospital. Patients requiring preoperative CT-guided localization and puncture will receive an ultrasound-guided deep SCTL block (T group) or superficial SCTL block (S group) 30 minutes before the procedure, with 10 patients in each group. The block sites will be at the surgical side T4 and T6 levels, using 20 mL of a nerve block solution containing 0.375% ropivacaine mixed with 2 mL of iohexol (total 20 mL).

Following the nerve block, patients will be placed in the supine position, and after 30 minutes, a blinded investigator will assess sensory loss using cold stimulation at the anterior chest wall (midclavicular line), lateral chest wall (posterior axillary line), and posterior chest wall (paravertebral region). Subsequently, patients will undergo routine CT-guided lesion localization and 3D imaging technology will be used to evaluate drug diffusion patterns for the two block techniques.

Any adverse events occurring during the trial will be managed according to the study protocol and recorded accordingly.

DETAILED DESCRIPTION:
Thoracoscopic lobectomy is a commonly performed surgical procedure known for its minimal invasiveness and rapid recovery. Effective pain management during surgery is crucial for patient recovery and surgical outcomes. To further enhance postoperative comfort and accelerate recovery, the combined use of general anesthesia and regional blockade techniques has been increasingly recommended in recent years. Regional blockade not only effectively alleviates postoperative pain but also helps reduce the consumption of general anesthetic agents, facilitating faster recovery.

Thoracic paravertebral block (TPVB) is an effective regional anesthesia technique that provides a novel option for postoperative pain management in thoracoscopic lobectomy. TPVB involves the injection of local anesthetics near the intervertebral foramen adjacent to the thoracic spinal nerves, achieving blockade of the ipsilateral thoracic somatic and sympathetic nerves. It is primarily used for postoperative analgesia in rib fractures, breast surgery, thoracotomy, and thoracoscopic procedures. To ensure the effectiveness of regional blockade and optimize surgical turnover time, TPVB is typically performed in the pre-anesthesia room 30 minutes before surgery. This approach maximizes its analgesic benefits and promotes rapid postoperative recovery.

With the advancement of ultrasound-guided nerve block techniques, the incidence of complications such as pneumothorax and hemothorax associated with TPVB has significantly decreased. However, performing TPVB before surgery not only blocks thoracic nerves but also affects the sympathetic nerves regulating cardiac function. Inhibition of the sympathetic nervous system can lead to reduced myocardial contractility and heart rate, along with decreased peripheral vascular resistance, thereby increasing the incidence of hypotension during general anesthesia induction. This remains a critical clinical issue requiring urgent resolution.

The thoracic paravertebral space is a wedge-shaped space located on both sides of the thoracic vertebrae. Its medial boundary consists of the vertebral body, intervertebral disc, and intervertebral foramen, which connect to the epidural space. The lateral boundary extends to the intercostal space, the anterior boundary is formed by the pleura, and the posterior boundary consists of the superior costal transverse ligament (SCTL). Within this space lie structures such as the intercostal arteries and veins, spinal nerve roots, dorsal branches of spinal nerves, intercostal nerves, communicating branches, sympathetic chain, and adipose tissue.

Costache et al. demonstrated through cadaveric dye injection studies that dye diffused within the thoracic paravertebral space, suggesting that it is not a completely enclosed anatomical compartment and that the SCTL does not act as a diffusion barrier for local anesthetics. Furthermore, Cho TH used micro-CT imaging to confirm that the thoracic paravertebral space is extremely narrow and that the SCTL does not form a closed posterior boundary. This finding indicates that drug injection on the superficial side of the SCTL can also spread into the thoracic paravertebral space.

Compared to conventional TPVB, injecting local anesthetics into the superficial layer of the SCTL allows the drugs to diffuse through the costotransverse ligament into the paravertebral space. With the same volume of local anesthetic, a smaller amount reaches the paravertebral space in a shorter time, resulting in a milder effect and less impact on sympathetic nerves. Theoretically, this approach may reduce the incidence of hypotension.

This study aims to investigate whether performing TPVB at the superficial layer of the SCTL (without puncturing through the ligament) provides more stable hemodynamics during anesthesia induction compared to the conventional deep approach (where the needle penetrates the SCTL), while maintaining equivalent analgesic effects for thoracoscopic lung resection surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for elective two-port video-assisted thoracoscopic lobectomy
* Age: ≥18 years
* ASA classification: I-III
* BMI: 18-30 kg/m²

Exclusion Criteria:

* Severe hypertension (SBP ≥180 mmHg or DBP ≥110 mmHg)
* MAP <70 mmHg before anesthesia induction
* Emergency surgery
* Severe cardiovascular disease, including history of cerebral or thoracic/abdominal aortic aneurysm
* Congestive heart failure (New York Heart Association class III or IV)
* Untreated or unstable ischemic heart disease
* Severe aortic or mitral valve disease
* Pregnancy or lactation
* Coagulation disorders
* Bacteremia, sepsis, or infection at the puncture site
* Allergy to study-related drugs
* Severe liver and kidney dysfunction
* Neurological disorders, spinal disease (deformity or trauma), history of spinal surgery, or abnormal skin sensation in the thoracic or back region
* Existing or anticipated difficult airway management
* Other conditions deemed unsuitable for inclusion by the investigators Forty patients who required CT (3D) imaging technology to observe drug diffusion after the implementation of the two methods were included as follows: patients who were scheduled to undergo double-hole thoracoscopic lobectomy, aged ≥18 years, ASA grade I to III, BMI 18 to 30kg/m2, and required preoperative CT localization. Exclusion criteria In addition to the above conditions, patients with a history of anaphylaxis induced by contrast agents should be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 168 (Estimated)
Dates: Start 2025-05-25 (Estimated); Primary Completion 2026-06-25 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of hypotension | From the beginning of induction to 5 minutes after induction
  Incidence of hypotension during the induction period of general anesthesia (from the beginning of induction to 5 minutes after induction).Definition of hypotension: a 20% decrease in MAP or a MAP absolute value < 65 mmHg during this period.

SECONDARY OUTCOMES:
Incidence of severe hypotension | From the beginning of induction to 5 minutes after induction
  The incidence of severe hypotension during the induction period of general anesthesia (from the beginning of induction to 5 minutes after induction). Definition of severe hypotension: a 30% decrease in MAP or a MAP absolute value < 55 mmHg.
VAS scores | 4 and 24 hours after surgery
  The Visual Analog Scale (VAS) is used for assessing pain intensity. It consists of a continuous 10 cm (or 100 mm) line on which patients indicate their perceived level of pain or another symptom by marking a point along the scale.
  VAS Scale Minimum and Maximum Values Minimum value (0 cm or 0 mm): This represents no pain or the least possible intensity of the measured symptom.
  Maximum value (10 cm or 100 mm): Represents the worst imaginable pain or the most severe intensity of the measured symptom.
  Interpretation of Higher Scores Higher VAS scores indicate worse outcomes, meaning greater pain intensity or more severe symptoms.
  Lower VAS scores indicate better outcomes, meaning less pain or milder symptoms.
  Common VAS Score Ranges for Pain
  Pain levels are often categorized as follows:
  0 mm: No pain 1-3 mm: Mild pain 4-6 mm: Moderate pain 7-10 mm: Severe pain
HR values | Intraoperative
  HR values were recorded before the block, during induction (per minute), and when hypotension occurred.
MAP values | Intraoperative
  MAP values were recorded before the block, during induction (per minute), and when hypotension occurred.
SV values | Intraoperative
  SV values were recorded before the block, during induction (per minute), and when hypotension occurred.
CI values | Intraoperative
  CI values were recorded before the block, during induction (per minute), and when hypotension occurred.
Use of vasoactive drugs | From the beginning of induction to 5 minutes after induction
  Record the use of vasoactive drugs during induction.
Use of propofol and remifentanil | Anesthesia induction and during operation
  The amount of propofol and remifentanil used during operation and anesthesia induction were recorded
Surgery duration | Intraoperative
  Surgery duration was recorded from skin incision to wound closure, measured in minutes.
Puncture related adverse events | Recorded during the operation
  Records of puncture-related adverse events (whether hemothorax, pneumothorax, local hematoma, local anesthetic poisoning, epidural block, or general spinal anesthesia).
Score of QOR-15 | 24 hours after surgery
  The QOR-15 score 24 hours after operation was recorded
The use of analgesic pump and additional analgesic drugs | 24 hours after surgery
  The use of analgesic pump (oxycodone dosage, first compression time, effective compression times, actual compression times) and the use of additional analgesic drugs were recorded within 24 hours.
Puncture-related complications | 72 hours after surgery
  The puncture-related complications were observed within 72 hours after the operation.
Satisfaction survey | 72 hours after surgery
  The satisfaction survey of patients was recorded 72 hours after the operation
Intraoperative intravenous infusion volume | Intraoperative
  Intraoperative intravenous (IV) infusion volume refers to the total amount of fluids administered intravenously during surgery.
Intraoperative urine volume | Intraoperative
  Intraoperative urine volume refers to the amount of urine output measured during surgery.
Intraoperative blood loss | Intraoperative
  Typically measured in milliliters (mL). Estimated using: Suction canister volume (after subtracting irrigation fluids). Surgical sponges and gauze weighing (1g weight increase ≈ 1mL blood loss). Visual estimation by the surgical team.
Extubation time | up to 1 hour
  Extubation time refers to the time from the end of surgery to the removal of the endotracheal tube after general anesthesia.
CT (3D) imaging | 30 minutes after nerve block
  CT (3D) imaging was used to observe drug diffusion 30min after nerve block and cold stimulation was used to assess the degree of sensory loss, including the anterior chest wall (midclavicular line), lateral chest wall (posterior axillary line), and posterior chest wall (paravertebral area).

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoliang Wang, Study Director — The First Affiliated Hospital with Nanjing Medical University
Locations (1):
- Nanjing First Hospital, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No
In order to protect the privacy of participants, researchers decided not to make the data public. To obtain relevant data, researchers can be contacted if necessary.